CLINICAL TRIAL: NCT02410785
Title: Efficacy of Polyglucosamine for Weight Loss - in a Randomized, Double-blind, Placebo-controlled Clinical Investigation
Brief Title: Efficacy of Polyglucosamine for Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Certmedica International GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 001/09; U1111-1123-0658 (Other: WHO)
Record Dates: First submitted 2015-03-27; First posted 2015-04-08 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2015-03

CONDITIONS: Overweight and Obesity
Keywords: obesity,; body weight,; overweight,; weight loss,; polyglucosamine,; L112; caloric restriction; physical activity
MeSH Terms: conditions — Overweight; Obesity; Body Weight; Weight Loss; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medical device polyglucosamine (Active Comparator): 2 times daily 2 tablets with the two main meals with the highest fat content. Participants follow the German guideline with a hypo-caloric (-500 kcal daily) lifestyle and increased physical activity.
  Interventions: Device: Polyglucosamine
- Placebo (Placebo Comparator): 2 times daily 2 tablets with the two main meals with the highest fat content. Participants follow the German guideline with a hypo-caloric (-500 kcal daily) lifestyle and increased physical activity.
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Polyglucosamine — ß-1,4 polymer of D-glucosamine and N-acetyl-D-glucosamine from the shells of crustaceans
  Arms: Medical device polyglucosamine
Other: Placebo — Placebo tablet
  Arms: Placebo

SUMMARY:
The polyglucosamine, specification L112 is a medical device and in this clinical trial used for weight reduction of overweight and obese participants. The rationale for this study is to show that overweight can be reduced by taking 2 times daily 2 tablets with the main meals with the highest fat content.

DETAILED DESCRIPTION:
To have a comparable diet condition, all participants in both groups had to follow the recommendations of the German clinical practice guidelines on the management and prevention of obesity.

One group had to take the polyglucosamine tablets and the other group placebo tablets for at least 24 weeks. It is known, that polyglucosamine is a fat binder acting in a physical-chemical manner, the positive charged fiber is bound to the negative charged dietary fat and this complex in unable to pass the gut wall into the body but is naturally excreted, hence this energy is not available. Therefore, this medical device should show a measurable reduction in body weight.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 26 and < 45
* waist circumference of more than 88 cm for women and greater than 102 for men.

Exclusion Criteria:

* pregnancy or breast-feeding, alcohol abuse, drug abuse or drug addiction, inability to fulfill the criteria of the trial protocol, cancer diseases, malignant tumors, pre-existence of chronic intestinal disease and known hypersensitivity reactions to crustaceans

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2009-08; Primary Completion 2009-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Number of participants who could reduce their body weight by 5 or more per cent compared to the initial body weight. | 24 weeks

SECONDARY OUTCOMES:
Change of body weight in kg | 24 weeks
Change of BMI | 24 weeks
Reduction of waist circumference | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karina Pokhis, MD, Principal Investigator — Salztal Klinik GmbH
Locations (2):
- Salztal Klinik GmbH, Bad Soden-Salmünster, Hessia, Germany
- MAP Center, Rende, Cosenza, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pokhis K, Bitterlich N, Cornelli U, Cassano G. Efficacy of polyglucosamine for weight loss-confirmed in a randomized double-blind, placebo-controlled clinical investigation. BMC Obes. 2015 Jun 10;2:25. doi: 10.1186/s40608-015-0053-5. eCollection 2015. PMID 26217540